CLINICAL TRIAL: NCT01034033
Title: Genetic & Pathological Studies of BRCA1/BRCA2: Associated Tumors & Blood Samples
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Breast Cancer Research Foundation (Other); Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-11872; SU-11022007-786 (Other: Stanford University); BRSNSTU0020 (Other: OnCore)
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Ovarian Cancer; Gynecologic Cancers; Ovarian/Peritoneal/Fallopian Cancer
Keywords: quality of life
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and breast tissues
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to try to understand the biology of development of breast, ovarian, fallopian tube, peritoneal or endometrial cancer from persons at high genetic risk for these diseases. The influence of environmental factors on cancer development in individuals and families will be studied. The efficacy of treatments for these diseases will be evaluated.

DETAILED DESCRIPTION:
1. To establish a demographic database to evaluate the efficacy of medical interventions in patients and relatives who carry BRCA1 and 2 mutations and to compare these outcomes to patients who do not carry a BRCA1 or 2 mutation.
2. To obtain blood samples from patients who undergo genetic testing to a) evaluate the incidence of genetic modifier polymorphisms involved in the development of cancer in BRCA1 and 2 mutation carriers and to compare this incidence to non-BRCA 1 and 2 carriers. b) to understand the interaction of genetic modifiers and BRCA1 and 2 in the development of cancer. c) to determine the effect of environmental influences on the incidence of polymorphisms in genetic modifiers and on the penetrance of BRCA1 and 2 mutations by linking information from our demographic database to blood samples and
3. To obtain tumor tissue from BRCA1 and 2 carriers to utilize for gene expression studies.
4. To establish a cohort of sporadic breast cancer patients, or women with no family history of cancer in a first degree relative, to serve as a comparison group to women with strong family history of breast cancer.
5. To establish a cohort of healthy volunteers without personal or family history of cancer to serve as a comparison group to women with sporadic and familial breast cancer.

ELIGIBILITY:
Inclusion Criteria:

I. Women who have a high risk of developing breast or ovarian cancer due to a known germline mutation in the BRCA1/2, PTEN, CDH1, or TP53 cancer susceptibility genes, or due to strong family history of either breast or ovarian cancer, in the absence of known cancer susceptibility gene mutation.

II. Women who are approaching surgery for resection of a pelvic mass, which is considered suspicious for neoplasia by radiologic or clinical criteria; such women may or may not also meet criteria for inclusion in group I.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women who have a high risk of developing breast or ovarian cancer due to a known germline mutation in the BRCA1/2, PTEN, CDH1, or TP53 cancer susceptibility genes, or due to strong family history of either breast or ovarian cancer, in the absence of known cancer susceptibility gene mutation.
Sampling Method: Non-Probability Sample
Enrollment: 3300 (Estimated)
Dates: Start 2001-08; Primary Completion 2099-01 (Estimated); Study Completion 2099-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James M Ford, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No